CLINICAL TRIAL: NCT02824549
Title: An Evaluation of the Usability, Skin Reactions and Accuracy of the FreeStyle Libre Flash Glucose Monitoring System
Brief Title: An Evaluation of the FreeStyle Flash Glucose Monitoring System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Ingrid Arijs, Prof. dr. G. Massa, MD, PhD - Pediatric Endocrinologist, Jessa Hospital
Other Study IDs: B243201628915
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-07

CONDITIONS: Flash Glucose Monitoring; Skin Reactions
Keywords: Flash glucose monitoring; skin reactions; usability; accuracy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: FreeStyle Libre Flash Glucose Monitoring

SUMMARY:
The usability, skin reactions and accuracy of the FreeStyle Libre glucose monitoring system in children will be evaluated by questionnaires, pictures of the insertion site and comparison of the glucose results with capillary blood glucose determinations.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes mellitus
* being followed in the Pediatric Diabetes Unit of the Jessa Ziekenhuis

Exclusion Criteria:

-

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with type 1 diabetes mellitis using the FreeStyle Libre Flash glucose monitoring system
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Usability of the FreeStyle glucose monitoring systeem | 0.5 year follow-up
  The usability will be evaluated by a short questionnaire.

SECONDARY OUTCOMES:
Skin reactions to the sensor : e.g. allergic reaction, red mark, blister | 0.5 year follow-up
  The skin reactions will be evaluated by a questionnaire and a picture will be taken when skin reactions are present.
Accuracy of the FreeStyle Libre glucose monitoring system | 0.5 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Guy Massa, MD, PhD, Study Director — Department of Pediatric Diabetology, Jessa Ziekenhuis, Stadsomvaart 11, B3500 Hasselt, Belgium; Renate Zeevaert, MD, PhD, Principal Investigator — Department of Pediatric Diabetology, Jessa Ziekenhuis, Stadsomvaart 11, B3500 Hasselt, Belgium
Locations (1):
- Jessa Hospital, Hasselt, Belgium